CLINICAL TRIAL: NCT00818831
Title: Phase I Safety and Pharmacokinetic Study of QBI-139 Injection Administered by Weekly Intravenous Infusion in Patients With Refractory Malignancies
Brief Title: A Study of QBI-139 in Subjects With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Quintessence Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: QBI-139 -101; CO 08912 (Other: University of Wisconsin Comprehensive Cancer Center); 2009-0716 (Other: MD Anderson)
Record Dates: First submitted 2009-01-07; First posted 2009-01-08 (Estimated); Last update posted 2015-01-28 (Estimated); Status verified 2015-01

CONDITIONS: Solid Tumors
Keywords: Advanced, refractory solid tumors

INTERVENTIONS:
Drug: QBI-139 — QBI-139 is being administered once a week over a two hour infusion in escalating doses.

SUMMARY:
The purposes of this trial are:

* To evaluate the toxicity and tolerability of QBI-139 in patients with advanced refractory solid tumors.
* To determine the maximum tolerated dose of QBI-139 in patients with advanced, refractory solid tumors.

Patients will receive QBI-139 by IV infusion over at least one hour once weekly for three weeks. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3 to 6 patients receive escalating doses of QBI-139 until the maximum tolerated dose (MTD) is determined.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be refractory to or intolerant of established therapy known to provide clinical benefit for their condition, i.e., patients must not be candidates for regimens known to provide clinical benefit.
* Patients must have measurable (as defined by Response Evaluation Criteria in Solid Tumors (RECIST) criteria) solid tumors.
* Prior chemotherapy and radiation therapy are allowed (at least 4 weeks must have passed from prior chemotherapy and radiotherapy (6 weeks for nitrosoureas or mitomycin C)), provided that clinically significant toxicity related to prior chemotherapy or radiotherapy has returned to baseline or National Cancer Institute (NCI) Common Toxicity and Adverse Events (CTCAE) grade ≤ 2 and are not expected to recover further. The toxicities specifically exclude alopecia.
* Age >18 years.
* ECOG performance status <2.
* Life expectancy of greater than 12 weeks, as estimated by Principal Investigator.
* Patients must have normal organ and marrow function as defined in the protocol.
* The effects of QBI-139 on the developing human fetus are unknown. Therefore, both men and women should not attempt to conceive and women should not be pregnant or breast-feeding while taking part in this study (or for 90 days after completing the study).
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Concurrent treatment with an investigational agent other than the investigational agent(s) used in this study OR treatment within 4 weeks of study entry with any investigational agent(s) or device(s).
* Failure to recover fully (as judged by the Investigator) from prior surgical procedures.
* Patients with known brain metastases or leptomeningeal carcinomatosis
* Patients who have had a gastrointestinal bleed requiring transfusion within the past 6 months or active Grade 2 or higher diarrhea
* Treatment with Ranpirnase (Onconase®)
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Women who are pregnant or breastfeeding
* Patients known to have HIV are ineligible
* Patients with known immunocompromised status or organ transplants will be excluded
* Patients must not have:

  * unstable angina (anginal symptoms at rest) within the past 6 months or
  * myocardial infarction within the past 6 months or
  * new onset angina within the last 3 months.
* QT prolongation (defined as QTc >450 msec for males and QTc >470 msec for females)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-01; Primary Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
To evaluate the toxicity and tolerability of and the maximum tolerated dose for QBI-139 in patients with advanced refractory solid tumors. | Cycle 1 (three weeks)

SECONDARY OUTCOMES:
To determine the patient response rate to QBI-139 using the RECIST criteria. | Duration of drug administration
To evaluate the pharmacokinetics of QBI-139 | Cycles 1 and 2 (six weeks)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - The University of Texas M. D. Anderson Cancer Center, Houston, Texas
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin

REFERENCES:
- See also: UW Carbone Cancer Clinical Trials webpage — http://www.uwhealth.org/onlineservices/cancertrials/
- See also: Phase I Clinical Trials Program at MD Anderson — http://www.mdanderson.org/education-and-research/departments-programs-and-labs/departments-and-divisions/investigational-cancer-therapeutics/index.html